CLINICAL TRIAL: NCT00573040
Title: Radiotherapy for Stage I-III Non-small Cell Lung Cancer to an Individualized MLD
Brief Title: Radiotherapy for NSCLC to a Individualized MLD
Acronym: BRONC MLD
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: MAASTRO clinic, MAASTRO clinic
Other Study IDs: BRONC MLD
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Radiotherapy; NSCLC; Stage III non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Inclusion criteria
  * Histological or cytological proven NSCLC
  * UICC stage I-III
  * Performance status 0-2
  * FeV1 and DLCO at least 30% of age-predicted value
  Exclusion criteria:
  * Not NSCLC or mixed NSCLC and other histologies (e.g. small cell carcinoma)
  * Stage IV
  * Performance status 3 or more
  * FeV 1 or DLCO < 30% of the age-predicted value

SUMMARY:
Our group has shown in a modeling study that increasing the radiation dose to pre-specified normal tissue dose constrains could lead to increased TCP with the same NTCP. In a subsequent phase I trial, the investigators showed the safety of this approach. Here, the investigators want to investigate its efficacy in a prospective study in patients with stage I-III NSCLC, who are selected for radical radiotherapy

DETAILED DESCRIPTION:
Eligible patients (see below) will receive radiotherapy to the primary tumor and the initially involved mediastinal lymph nodes to the following MLD (Mean Lung Dose):

* MLD=19 Gy when Fev1 and DLCO > 50% of the predicted value
* MLD=15 Gy when Fev1 and/or DLCO 40-49% of the predicted value
* MLD=10 Gy when Fev1 and/or DLCO <40% of the predicted value

Other dose-constrains: spinal cord max: 54 Gy, brachial plexus (Dmax):66 Gy Minimum tumor dose:79.2 Gy.

Radiotherapy will be delivered in twice-daily fractions of 1.8 Gy with 8 to 10 h as interfraction-interval, 5 days per week.

The radiation doses will be specified according to ICRU 50. Lung density corrections will be applied, as well as all standard QA procedures. Technical requirements are the same as in standard practice at MAASTRO clinic.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proven NSCLC
* UICC stage I-III
* Performance status 0-2
* FeV 1 and DLCO at least 30% of the age-predicted value

Exclusion Criteria:

* Not NSCLC or mixed NSCLC and other histologies (e.g. small cell carcinoma)
* UICC stage IV
* Performance status 3 or more
* FeV 1 and DLCO < 30% of the age-predicted value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Histological or cytological proven NSCLC
  * UICC stage I-III
  * Performance status 0-2
  * FeV 1 and DLCO at least 30% of the age-predicted value
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2005-08; Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
death | 2,3 and 5 years

SECONDARY OUTCOMES:
-progression-free interval -Dyspnea (CTCAE 3.0) -Dysphagia (CTCAE 3.0) -Patterns of recurrence | 2,3 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ruysscher, MD,PhD, Principal Investigator — MAASTRO clinic, Maastricht Radiation Oncology
Locations (1):
- MAASTRO clinic, Maastricht Radiation Oncology, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Nalbantov G, Kietselaer B, Vandecasteele K, Oberije C, Berbee M, Troost E, Dingemans AM, van Baardwijk A, Smits K, Dekker A, Bussink J, De Ruysscher D, Lievens Y, Lambin P. Cardiac comorbidity is an independent risk factor for radiation-induced lung toxicity in lung cancer patients. Radiother Oncol. 2013 Oct;109(1):100-6. doi: 10.1016/j.radonc.2013.08.035. Epub 2013 Sep 14. PMID 24044794
- [Derived] Dehing-Oberije C, Aerts H, Yu S, De Ruysscher D, Menheere P, Hilvo M, van der Weide H, Rao B, Lambin P. Development and validation of a prognostic model using blood biomarker information for prediction of survival of non-small-cell lung cancer patients treated with combined chemotherapy and radiation or radiotherapy alone (NCT00181519, NCT00573040, and NCT00572325). Int J Radiat Oncol Biol Phys. 2011 Oct 1;81(2):360-8. doi: 10.1016/j.ijrobp.2010.06.011. Epub 2010 Oct 1. PMID 20888135